CLINICAL TRIAL: NCT06649305
Title: A Prospective Multicenter Clinical Study：IntracOnary neaR-Infrared Spectroscopy and OptIcal Coherence Tomography for Evaluating Coronary vulNerable Plaque in Patients With diabeTes
Brief Title: A Prospective Multicenter Clinical Study： IntracOronary neaR-Infrared Spectroscopy and OptIcal Coherence Tomography for Evaluating Coronary vulNerable Plaque in Patients With diabeTes
Status: Recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ORIENT
Record Dates: First submitted 2024-10-17; First posted 2024-10-18 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Coronary Heart Disease (CHD); Diabetes (DM)
Keywords: near-infrared spectroscopy
MeSH Terms: conditions — Coronary Disease; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental group: NIRS-OCT examination

SUMMARY:
To evaluate the correlation between maxLCBI4mm/FCTmin(a new index of lipid plaque based on NIRS-OCT technology) and fiber cap thickness , and the prognosis of patients, providing a new quantitative index for early, accurate and comprehensive identification of vulnerable plaques, and exploring preventive measures for adverse events such as cardiac death and recurrent myocardial infarction caused by vulnerable plaques, so as to improve the long-term prognosis of patients.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old or older, gender is not limited
2. Patients with diabetes who require an OCT examination or treatment under OCT guidance (diabetes definition: active treatment with insulin or oral hypoglycemic agents at admission). For patients with diabetes who are treated with diet only, abnormal fasting blood sugar (>7 mmol/l), blood sugar >11.1 mmol/l at any time, or abnormal glucose tolerance tests based on World Health Organization standards need to be recorded.
3. Be able to understand the purpose of clinical research, voluntarily participate can complete the observation as required and sign the informed consent form

5: Lesion stenosis greater than or equal to 50% without interventional treatment

6: The diameter of the blood vessel in the diseased segment is greater than or equal to 2.5 mm

Exclusion Criteria:

* 1: Severe coagulation dysfunction (APTT greater than 3 times the upper limit of the normal range)

  2: Severe hemodynamic disorder or shock that cannot be corrected

  3: Patients with renal impairment（eGFR<30 mL/min/1.73m2）

  4: Severe symptoms of heart failure (NYHA III and above) or left ventricular ejection fraction <30%

  5: The presence or suspected presence of infective endocarditis or systemic active infection

  6: Patients with refractory ventricular arrhythmias who have previously undergone coronary bypass transplantation (CABG) or plan to undergo CABG during the study

  7: Patients with serious concurrent diseases such as advanced cancer have a life expectancy of less than 24 months

  8: Pregnant or lactating women, have a family plan within 24 months or are unwilling to take effective contraceptive measures

  9: The target vessel has severe calcification or severe tortuosity, which cannot be examined by OCT

  10: Have participated in other clinical trials or are participating in other drug/device clinical trials within 3 months prior to enrollment and have not met the primary endpoint

  11: Investigators believe that those who are unnecessary for OCT or not suitable for inclusion in this trial.

  12: There are multiple lesions in the same blood vessel, and the non-target lesion distance requiring treatment vascular segment is less than 5mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years old or older ，with diabetes requiring an OCT examination or treatment under OCT guidance
Sampling Method: Non-Probability Sample
Enrollment: 1516 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2027-07-15 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
MACE events in the 24 months after operation | 24 months after operation
  record the MACE events (cardiac death, myocardial infarction, progressive angina, revascularization) after operation in 24 months

SECONDARY OUTCOMES:
The maxLCBI4mm/FCTmin ratio | 24 months after operation
  The maxLCBI4mm/FCTmin ratio is higher than 400/75
The maxLCBI4mm/FCTmin ratio | 24 months after operation
  The maxLCBI4mm/FCTmin ratio can be used as a continuous indicator

OTHER OUTCOMES:
Correlation between maxLCBI1mm and MACE events | 24 months after operation
  The association of maxLCBI1mm(the maximum lipid core load index in any 1mm long range as assessed by NIRS) with MACE events
Correlation between maxLCBI4mm and MACE events | 24 months after operation
Correlation between the ratio of maxLCBI1mm to the thinnest fiber cap thickness with MACE events | 24 months after operation
The newly defined vulnerable plaque 1) Presence of minimum lumen area <3.5 mm² 2) maxLCBI4mm / FCTmin higher than the median | 24 months after operation
  The newly defined vulnerable plaque is more likely to be the primary culprit for MACE events than the traditionally defined vulnerable plaque
Correlation between D-LCBI4mm lipid core load index and MACE events | 24 months after operation

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided